CLINICAL TRIAL: NCT07337902
Title: Acetaminophen Versus Ibuprofen for Discomfort in Crohn's Disease (AVID-CD): An Open-Label Randomized Pilot Trial
Brief Title: Comparing Over the Counter Pain Medicines for Discomfort in Crohn's Disease (AVID-CD)
Acronym: AVID-CD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-2940
Record Dates: First submitted 2025-12-19; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Crohn's Disease (CD); Dysmenorrhea Primary
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acetaminophen, Ibuprofen, Acetaminophen, Ibuprofen (Experimental): Participants will receive medications for each of four menstrual cycles in the following order: 1. Acetaminophen 2. Ibuprofen 3. Acetaminophen 4. Ibuprofen
  Interventions: Other: Acetaminophen; Other: Ibuprofen
- Acetaminophen, Ibuprofen, Ibuprofen, Acetaminophen (Experimental): Participants will receive medications for each of four menstrual cycles in the following order: 1. Acetaminophen 2. Ibuprofen 3. Ibuprofen 4. Acetaminophen
  Interventions: Other: Acetaminophen; Other: Ibuprofen
- Ibuprofen, Acetaminophen, Ibuprofen, Acetaminophen (Experimental): Participants will receive medications for each of four menstrual cycles in the following order: 1. Ibuprofen 2. Acetaminophen 3. Ibuprofen 4. Acetaminophen
  Interventions: Other: Acetaminophen; Other: Ibuprofen
- Ibuprofen, Acetaminophen, Acetaminophen, Ibuprofen (Experimental): Participants will receive medications for each of four menstrual cycles in the following order: 1. Ibuprofen 2. Acetaminophen 3. Acetaminophen 4. Ibuprofen
  Interventions: Other: Acetaminophen; Other: Ibuprofen

INTERVENTIONS:
Other: Acetaminophen — Participants will receive oral acetaminophen 650 mg three times daily for three days during two of four menstrual cycles by random assignment at the onset of cramps.
  Other Names: Tylenol
Other: Ibuprofen — Participants will receive oral ibuprofen 400 mg three times daily for three days during two of four menstrual cycles by random assignment at the onset of cramps.
  Other Names: Advil

SUMMARY:
The purpose of this pilot study is to prepare for a larger study that will compare the effectiveness and safety of two common pain medications, ibuprofen and acetaminophen, to help treat period cramps in women with Crohn's disease. The goal of this study is to identify any challenges in running a larger study. The investigators will track how many people sign up for the study, how well participants follow the study plan, how many people stay in the study, and whether they are able to complete all the study activities, such as taking the medication, submitting samples, and filling out surveys.

During the study, participants will undergo a screening visit that includes a blood draw, physical exam, pregnancy test, stool testing, and complete surveys about Crohn's disease and menstrual cycles. Once this visit is complete, the rest of the study will occur at home.

Participants will be assigned to take either ibuprofen or acetaminophen to help treat period cramps for four menstrual cycles in a row. Participants will take ibuprofen for two cycles and acetaminophen for two cycles. Participants will know which medication is being taken at any given time, but the order in which they take the medications will be randomly assigned.

Before each menstrual cycle, participants will submit a stool sample and fill out a short (<1 minute) electronic survey. When participants develop period cramps, they will take the assigned medication for three days and fill out short (<1 minute) electronic surveys about their cramps. After participants finish taking the medication for three days, they will submit another stool sample and fill out two more short (<1 minute) electronic surveys. After have completing this process for four menstrual cycles, a remote interview with a researcher to give feedback on the study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-44 years
* Assigned female at birth
* Crohn's Disease (CD) diagnosis
* In stable clinical remission from CD, defined as a short Crohn's Disease Activity Index (CDAI; See Table 3) <150 without use of corticosteroids
* Self-reported primary dysmenorrhea
* Regular menstrual cycles occurring every 23-35 days
* Using an appropriate contraceptive method or abstinence

Exclusion Criteria:

* Any of the following conditions: endometriosis, adenomyosis, polycystic ovarian syndrome, endometrial fibroids/polyps, chronic pelvic inflammatory disease, a history of pelvic surgery including hysterectomy, any other pathological pelvic conditions, or current pregnancy
* Plans to become pregnant during the study period
* Use of an oral contraceptive for less than 3 months, on an unstable oral contraceptive dose within the last 3 months, switched from one oral contraceptive to another within the last 3 months or intend to do so during the course of the trial
* Taking hormone therapy including estrogen or progesterone that is not part of a hormonal contraceptive
* Known hypersensitivity or contraindication to ibuprofen or acetaminophen
* Inability to complete REDCap questionnaires (including confusion despite training and/or lack of smart phone and/or computer access).
* Not able to speak and read English language.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Who Express Interest in the Study Out of Those Contacted | from first contact to informed consent, up to 2 years
  Accrual will be determined as the proportion of participants who express interest in the study out of those contacted
Proportion of participants who enroll out of those who expressed interest in the study | from first contact to informed consent, up to 2 years
  Accrual will be determined by the proportion of participants who enroll out of those who expressed interest in the study
Proportion of participants who meet the minimum adherence needed to contribute effectively to a subsequent study out of those randomized | enrollment to completion of study, approximately 2.5 years
  Protocol Adherence will be determined by the proportion of participants who meet the minimum adherence needed to contribute effectively to a subsequent study out of those randomized

SECONDARY OUTCOMES:
Number of Participants who meet exclusion criteria out ot the Total Screened | first recruitment through screening, approximately 2 years
  Recruitment Barriers will be determined among screened participants by the number who meet exclusion criteria
Reasons for Declining Study Participation by Category | first contact through screening, approximately 2 years
  Recruitment Barriers will be summarized by the number of participants among those eligible who have been screened listed by reason(s) for declining participation.
Number of Participants who consented that do not complete baseline visit | first contact through end of study, approximately 2 years
  Recruitment Barriers will be summarized as the number of participants who consented that do not complete baseline visit
Number of subjects who return all stool samples | enrollment through end of study, approximately 5 months
  Adherence Rates will be summarized as the number of subjects who return all stool samples
Number of participants who take the study drugs per protocol | enrollment through end of study, approximately 5 months
  Adherence Rates will be summarized by the number of participants who take the study drugs per protocol
Number of participants who complete the dysmenorrhea surveys | enrollment through end of study, approximately 5 months
  Adherence rates will be summarized by the number of participants who complete the dysmenorrhea surveys
Number of subjects who complete the Irritable Bowel Syndrome (IBD) surveys | enrollment through end of study, approximately 5 months
  Adherence Rates will be summarized by the number of subjects who complete the Irritable Bowel Syndrome (IBD) surveys
Number of subjects who complete all study activities per protocol | enrollment through end of study, approximately 5 months
  Adherence rates will be summarized by the number of subjects who complete all study activities per protocol
Number of participants who delay participation due to lack of dysmenorrhea | enrollment to end of study, approximately 5 months
  Adherence barriers will be summarized by the number of participants who delay participation due to lack of dysmenorrhea
Number of participants who delay participation or drop out due to active IBD | enrollment to end of study, approximately 5 months
  Adherence Barriers will be summarized by the number of participants who delay participation or drop out due to active IBD
Number of participants who use study drug for other indications during the study | enrollment to end of study, approximately 5 months
  Adherence Barriers will be summarized by number of participants who use study drug for other indications during the study
Number of participants who use a rescue medication | enrollment to end of study, approximately 5 months
  Adherence Barriers will be summarized by number of participants who use a rescue medication
Reported barriers to compliance with procedures | following completion of fourth menstrual cycle, single interview lasting approximately one hour
  Participant qualitative interview feedback will be summarized by listing of reported barriers to compliance with procedures
Acceptability of study intervention and protocol | following completion of fourth menstrual cycle, single interview lasting approximately one hour
  Participant qualitative interview feedback will be summarized by number of participants reporting acceptability of study intervention and protocol
Areas of confusion regarding instructions or protocol | following completion of fourth menstrual cycle, single interview lasting approximately one hour
  Participant qualitative interview feedback will be summarized by a list of areas of confusion regarding instructions or protocol
Interest in stool bio-banking for future research | following completion of fourth menstrual cycle, single interview lasting approximately one hour
  Participant qualitative interview feedback will be summarized by number of subjects interested in stool bio-banking for future research

CONTACTS AND LOCATIONS:
Overall Officials: Erica J Brenner, MD, MSCR, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina.
Supporting Information: Study Protocol
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator who proposes to use the data has approved IRB, IEC, or REB and an executed data use/sharing agreement with the University of North Carolina.